CLINICAL TRIAL: NCT06917144
Title: Evaluating Repetitive Transcranial Magnetic Stimulation for Refractory Chronic Cluster Headache Prevention: Insights From a Randomised Crossover Pilot Trial
Brief Title: Refractory Chronic Cluster Headache: Exploring the Potential of Repetitive Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Javier Díaz de Terán, PhD, Instituto de Investigación Hospital Universitario La Paz
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PI-6581
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Refractory Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Other): The study consisted of two treatment periods (rTMS and sham stimulation), separated by a one-month washout period, and organized into two sequences (A and B)
  Sequence A:
  rTMS → washout → sham.
  Sequence B:
  sham → washout → rTMS.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Sham Stimulation
- Sequence B (Other): Sequence B:
  sham → washout → rTMS.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Sham Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Stimulation sessions were performed using a YINGCHI M-100 Ultimate device with liquid-cooled figure-8 coils.
  Patients attended 10-minute sessions daily for 10 consecutive working days. For rTMS, stimulation was delivered at an excitatory frequency of 10 Hz, targeting the M1, contralateral to the side of pain in the facial region.
  Each session consisted of the following steps.
  * 10 series: 60 pulses per series (600 pulses in total).
  * Rest intervals: 60 seconds between series.
  * Intensity: 70% of the resting motor threshold (RMT). RMT was determined using single-pulse stimulation over the M1 region controlling the abductor pollicis brevis muscle, localized via neuronavigation. The threshold was de-fined as the lowest stimulator intensity producing a motor-evoked potential amplitude >50 µV in at least 5 of 10 trials.
Device: Sham Stimulation — Sham Stimulation:
  The same device and protocol used for intervention protocol with Repetitive Transcranial Magnetic Stimulation were used for sham stimulation, but no active stimulation was delivered. The equipment produced identical sounds and appearances, thereby ensuring blinding.

SUMMARY:
The goal of this clinical trial is to learn if drug ABC works to treat severe asthma in adults. It will also learn about the safety of drug ABC. The main questions it aims to answer are:

Does Transcranial Magnetic Stimulation lower the number of attacks per week in patients with refractory cluster headache ?

Researchers will compare transcranial magnetic stimlation to a sham stimulation (a look-alike stimulation) to see if it works to prevent attacks of cluster headache.

Participants will:

Recieve stimulation for 10 minutes for 10 consecutive working days in 2 periods of time, separated by a 1 month washout period.

Visit the clinic for each treatment day. Keep a diary of their symptoms and the number of times they use a rescue medication

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with Chronic Cluster Headache (CCH) based on the International Classification of Headache Disorders 3rd Edition
* Diagnosed with refractory CCH based on the European Headache Federation criteria of 2014.

Exclusion Criteria:

* History of epilepsy.
* Concomitant diagnosis of any other headache (if the patient was unable to differentiate between them).
* Carriers of any electronic device, or any additional contraindication for Transcranial Magnetic Stimulation, such as pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Reduction in number of attacks per week | From enrollment to the end to follow up period, at 3 months after last treatment period (week 8)
  The mean change in the number of attacks per week at the end of each treatment period was compared with the baseline, from the time of informed consent until the last follow-up moment (3 months after the end of the second treatment period).

SECONDARY OUTCOMES:
Assessing the reduction in symptomatic medication use. | From enrollment to the end of follow up period, at 3 months after second treatment period (week 8)
  The use of symptomatic medication was assessed through electronic questionnaires completed by the patient.
  The mean change in the use of symptomatic medication at the end of each treatment period was compared with the baseline, from the time of informed consent until the last follow-up moment (3 months after the end of the second treatment period).
To assess the reduction in intensity of cluster headache attacks | From enrollment to the end of follow up period, at 3 months after second treatment period (week 8)
  The intensity of the attacks of cluster headache was assessed through electronic questionnaires completed by the patient, using the visual analogue scale from 1 to 10.
  The mean change in the intensity at the end of each treatment period was compared with the baseline, from the time of informed consent until the last follow-up moment (3 months after the end of the second treatment period).
To assess the change in duration in cluster headache attacks | From enrollment to the end of follow up period, at 3 months after second treatment period (week 8)
  The duration of the attacks of cluster headache was assessed through electronic questionnaires completed by the patient (minutes). The mean change in the duration at the end of each treatment period was compared with the baseline, from the time of informed consent until the last follow-up moment (3 months after the end of the second treatment period).
To assess the tolerability to treatment | From enrollment to the end of follow up period, at 3 months after second treatment period (week 8)
  The tolerability to treatment was assessed through electronic questionnaires completed by the patient, reporting any symptom experienced during treatment. It was then evaluated its possible relationship to rTMS. The adverse effects were evaluated from the time of informed consent until the last follow-up moment (3 months after the end of the second treatment period).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Portocarrero-Sanchez L, Rizea C, Diez-Tejedor E, Leon-Ruiz M, Diaz-de-Teran J. Evaluating Repetitive Transcranial Magnetic Stimulation for Refractory Chronic Cluster Headache Prevention: Insights from a Randomized Crossover Pilot Trial. Brain Sci. 2025 May 23;15(6):554. doi: 10.3390/brainsci15060554. PMID 40563725